CLINICAL TRIAL: NCT05561452
Title: The Efficacy of Single PRP Injection Compared With Placebo and Multiple PRP Injections in the Treatment of Rotator Cuff Syndrome: A Randomized Controlled Study
Brief Title: The Efficacy of PRP Injection in the Treatment of Rotator Cuff Syndrome
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Elshan Hasanov, Research assistant doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROTCUFFPRP2022
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Pain; Musculoskeletal Diseases; Rotator Cuff Tendinopathy; Rotator Cuff Syndrome
Keywords: Platelet rich plasma ( PRP); Subacromial injection; Rotator cuff tendinopathy; Rotator Cuff Syndrome
MeSH Terms: conditions — Shoulder Pain; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single PRP Injection + Exercise (Experimental): In single-PRP injection group, 10 ml of venous blood taken from the patients will be put into the T-LAB® PRP kit (T-Biotechnology Laboratory, İstanbul, Turkey) and will then be centrifuged at 3850 rpm for 8 minutes. Approximately 4 ml of the PRP obtained will be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. All injections will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote® My Lab 70 XVision 6-18 Mhz, linear probe).
  A home exercise program including Codman pendulum exercises, shoulder range of motion, stretching and strengthening exercises will be taught and the patients be instructed to perform at least for 20 minutes daily.
  Interventions: Other: Single PRP Injection
- Multiple PRP Injection+ Exercise (Experimental): In multiple-PRP injection group, two PRP injections will be performed with an interval of 3 weeks. 10 ml of venous blood taken from the patients will be put into the T-LAB® PRP kit (T-Biotechnology Laboratory, İstanbul, Turkey) and will then be centrifuged at 3850 rpm for 8 minutes. Approximately 4 ml of the PRP obtained will be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. All injections will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote® My Lab 70 XVision 6-18 Mhz, linear probe).
  A home exercise program including Codman pendulum exercises, shoulder range of motion, stretching and strengthening exercises will be taught and the patients be instructed to perform at least for 20 minutes daily.
  Interventions: Other: Multiple PRP Injections
- Saline Injection + Exercise (Sham Comparator): In placebo-injection group,10 ml of venous blood will be taken and after the same waiting time 4 ml of 0.9% saline will be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. All injections will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote® My Lab 70 XVision 6-18 Mhz, linear probe).
  A home exercise program including Codman pendulum exercises, shoulder range of motion, stretching and strengthening exercises will be taught and the patients be instructed to perform at least for 20 minutes daily.
  Interventions: Other: Placebo Injection

INTERVENTIONS:
Other: Single PRP Injection — In single-PRP injection group, 10 ml of venous blood taken from the patients will be put into the T-LAB® PRP kit (T-Biotechnology Laboratory, İstanbul, Turkey) and will then be centrifuged at 3850 rpm for 8 minutes. Approximately 4 ml of the PRP obtained will be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. All injections will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote My Lab 70 XVision 6-18 Mhz linear probe).
  A physical therapy program including Codman pendulum exercises, shoulder range of motion, stretching and strengthening exercises will be given and be performed at least for 20 minutes daily.
  Arms: Single PRP Injection + Exercise
Other: Multiple PRP Injections — In multiple-PRP injection group, two PRP injections will be performed with an interval of 3 weeks. 10 ml of venous blood taken from the patients will be put into the T-LAB® PRP kit (T-Biotechnology Laboratory, İstanbul, Turkey) and will then be centrifuged at 3850 rpm for 8 minutes. Approximately 4 ml of the PRP obtained is planned to be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. All injections will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote My Lab 70 XVision 6-18 Mhz linear probe).
  A physical therapy program including Codman pendulum exercises, shoulder range of motion, stretching and strengthening exercises will be given and be performed at least for 20 minutes daily.
  Arms: Multiple PRP Injection+ Exercise
Other: Placebo Injection — In placebo-injection group,10 ml of venous blood will be taken and after the same waiting time 4 ml of 0.9% saline will be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. All injections will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote My Lab 70 XVision 6-18 Mhz linear probe).
  A physical therapy program including Codman pendulum exercises, shoulder range of motion, stretching and strengthening exercises will be given and be performed at least for 20 minutes daily.
  Arms: Saline Injection + Exercise

SUMMARY:
The aim of this study is to investigate the efficacy of single PRP injection compared with placebo and multiple PRP injections on pain, quality of life, shoulder function and muscle strength in the treatment of patients who have tendinopathy and/or partial tear in the rotator cuff.

DETAILED DESCRIPTION:
The study is a prospective double-blind randomized placebo-controlled trial. The study population is consisted of patients aged 18-65 years, who applied to the Department of Physical Medicine and Rehabilitation, Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey and were diagnosed with rotator cuff tendinopathy and/or partial tear in the supraspinatus tendon (< %50) by clinical and MRI examination, and met the inclusion criteria. The patients will be randomized into 3 groups using a closed envelope method; 1) Single PRP injection, 2) Single placebo injection, and 3) Two PRP injections applied 3 weeks apart. All injections will be performed into the subacromial space under ultrasound guidance. The same physical therapy program will be given to all groups and will be performed at least for 20 minutes daily.

The randomization will be done using the closed envelope method by a researcher who will not perform injections nor evaluate the patients, and to provide blindness, the injectors to be used will be covered with non-transparent tapes by the same investigator. The patients, the physician to make the evaluations, and the physician to perform injections will be blinded to the groups. The solution to be injected will be prepared by another researcher who is not blind. PRP injections will be prepared as follows;10 ml of venous blood taken from the patients will be put into the T-LAB® PRP kit (T-Biotechnology Laboratory, İstanbul, Turkey). The obtained blood will then be centrifuged at 3850 rpm for 8 minutes. Approximately 4 ml of the PRP obtained will be injected into the subacromial space using the lateral subacromial injection method under ultrasound guidance. The same amount of blood will be taken for the placebo injection group and after the same waiting time 4 ml of 0.9% saline will be injected using the same method.

Ultrasound guided lateral subacromial injection method will be used. For a safer and more efficient injection, all applications will be performed in the sagittal axis with the long axis in-plane technique, using the ultrasound device (Esaote® My Lab 70 XVision 6-18 Mhz linear probe). To obtain an optimal subacromial appearance with shoulder ultrasonography (USG), the patients will sit upright with their arms back, internally rotated, shoulder hyperextended and elbow flexed to 90° and forearm parallel to the floor. USG in-plane technique will be used in the subacromial region to confirm that the needle stays in the correct place as it is advanced.

Shoulder range of motion will be measured. The level of pain at rest, during motion and during the night will be evaluated with the visual analog scale (VAS). Constant Murley scale and Shoulder Pain and Disability Index (SPADI) will be used for functional evaluation. Quality of life will be assessed with Short-Form 36 (SF-36). Upper extremity muscle strength will be measured with the Isomed-2000® isokinetic device.

The participants in single-PRP injection and single-Placebo injection groups will be evaluated before the injection and 4 and 12 weeks later. Those in the two PRP injections group will be evaluated before the first injection, and 4 and 12 weeks after the second injection.

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder pain for at least 6 weeks in the participants with 18-65 years of age
2. Positivity of shoulder impingement tests on examination (Neer test, Hawkins Kennedy test)
3. Findings related to rotator cuff tendinopathy and partial tear in the supraspinatus tendon (< 50%) on MRI

Exclusion Criteria:

1. Pregnancy
2. Inflammatory rheumatologic diseases
3. History of malignacy
4. Having received physical therapy and rehabilitation for the shoulder in the last 3 months
5. Local injection therapy to the shoulder in the last 6 months
6. History of trauma, surgery or fracture in the aching shoulder region in the last 6 months
7. Presence of osteoarthritis findings and labral pathologies, adhesive capsulitis, calcific tendinitis and full-thickness total rupture of the rotator cuff tendons on MRI.
8. Cervical radiculopathy
9. Cervical myofascial pain syndrome
10. Presence of cardiac pacemaker
11. Bleeding diathesis
12. Body implant with electronic or battery system
13. Acute infections
14. Tuberculosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | up to 12th week
  Pain intensity will be measured with Visual Analog Scale (VAS) for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity. The level of pain at rest, during motion and during the night will be evaluated with the visual analog scale (VAS). Changes from baseline VAS scores will be assessed at 4th and 12th weeks.

SECONDARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | up to 12th week
  Shoulder Pain and Disability Index (SPADI) is a two-part scale that evaluates pain and function.The first part questions pain, the second part questions disability. In the pain section consisting of 5 items, the pain felt during activities of daily living is measured using a 10-unit VAS, and in the disability section, the difficulty encountered during activities of daily living is measured througout 8-items. The score of both sections and the total score are calculated with a special formula. Changes from baseline SPADI will be assessed at 4th and 12th weeks.
The 36-item Short Form Health Survey（SF-36） | up to 12th week
  The Short Form 36 (SF-36) is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score is between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Higher scores indicate better quality of life related to health. Changes from baseline SF-36 scores will be assessed at 4th and 12th weeks.
Range of Motion（ROM） | up to 12th week
  Range of Motion（ROM）of the shoulder will be measured in 5 planes. It includes abduction in the frontal plane, forward flexion, extension, internal rotation and external rotation with the arm at 0° of abduction. Changes from baseline ROM scores will be assessed at 4th and 12th weeks.
Constant Murley Score (C-MS) | up to 12th week
  The Constant-Murley Shoulder Score (C-M Score) is a clinical and functional assessment scale that evaluates the functional status of a normal, diseased or treated shoulder. Comparisons can be made in pre-treatment and post-treatment follow-up. Evaluated parameters were pain (15 points), activities of daily living (20 points), ROM (40 points), and strength (25 points). Scoring that measures the functionality of the shoulder consists of 100 points in total. C-M score; It is classified as excellent (90-100), good (80-89), moderate (70-79) and poor (<70). Changes from baseline C-M scores will be assessed at 4th and 12th weeks.
Isokinetic Test | up to 12th week
  Isokinetic contraction is defined as contraction at a constant rate throughout the entire range of motion and at an equal rate at all angles of motion. No matter how hard a person moves the device, they can never exceed the predetermined speed (for example, 90 degrees per second). It is advantageous that the desired muscle or muscle groups can be evaluated in isolation and that the measurements are comparable. The isokinetic strength assessment of the patients during internal and external rotation of the shoulder will be made with an isokinetic device (IsoMed 2000, Isokinetic dynamometer, Germany). Measurements will be made by a physiotherapist with at least 5 years of device experience. Measurements will be made in 10 repetitions to increase reliability. Change from baseline upper extremity muscle strength with isokinetic device will be assessed at 4th and 12th weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Selma EROGLU, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahi̇sar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barreto RB, Azevedo AR, Gois MC, Freire MRM, Silva DS, Cardoso JC. Platelet-Rich Plasma and Corticosteroid in the Treatment of Rotator Cuff Impingement Syndrome: Randomized Clinical Trial. Rev Bras Ortop (Sao Paulo). 2019 Dec;54(6):636-643. doi: 10.1016/j.rboe.2018.03.002. Epub 2019 Dec 13. PMID 31875061
- [Background] Hurley ET, Hannon CP, Pauzenberger L, Fat DL, Moran CJ, Mullett H. Nonoperative Treatment of Rotator Cuff Disease With Platelet-Rich Plasma: A Systematic Review of Randomized Controlled Trials. Arthroscopy. 2019 May;35(5):1584-1591. doi: 10.1016/j.arthro.2018.10.115. Epub 2019 Apr 15. PMID 31000394
- [Background] Kim HM, Dahiya N, Teefey SA, Middleton WD, Stobbs G, Steger-May K, Yamaguchi K, Keener JD. Location and initiation of degenerative rotator cuff tears: an analysis of three hundred and sixty shoulders. J Bone Joint Surg Am. 2010 May;92(5):1088-96. doi: 10.2106/JBJS.I.00686. PMID 20439653
- [Background] Ozyalvac ON, Tuzuner T, Gurpinar T, Obut A, Acar B, Akman YE. Radiological and functional outcomes of ultrasound-guided PRP injections in intrasubstance meniscal degenerations. J Orthop Surg (Hong Kong). 2019 May-Aug;27(2):2309499019852779. doi: 10.1177/2309499019852779. PMID 31204581
- [Background] Vilchez-Cavazos F, Millan-Alanis JM, Blazquez-Saldana J, Alvarez-Villalobos N, Pena-Martinez VM, Acosta-Olivo CA, Simental-Mendia M. Comparison of the Clinical Effectiveness of Single Versus Multiple Injections of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2019 Dec 16;7(12):2325967119887116. doi: 10.1177/2325967119887116. eCollection 2019 Dec. PMID 31897409
- [Background] Walsh MR, Nelson BJ, Braman JP, Yonke B, Obermeier M, Raja A, Reams M. Platelet-rich plasma in fibrin matrix to augment rotator cuff repair: a prospective, single-blinded, randomized study with 2-year follow-up. J Shoulder Elbow Surg. 2018 Sep;27(9):1553-1563. doi: 10.1016/j.jse.2018.05.003. Epub 2018 Jul 9. PMID 29996980
- [Background] Kesikburun S, Tan AK, Yilmaz B, Yasar E, Yazicioglu K. Platelet-rich plasma injections in the treatment of chronic rotator cuff tendinopathy: a randomized controlled trial with 1-year follow-up. Am J Sports Med. 2013 Nov;41(11):2609-16. doi: 10.1177/0363546513496542. Epub 2013 Jul 26. PMID 23893418